CLINICAL TRIAL: NCT05875740
Title: Correlation of Memory CD8+ T Cells With Sepsis Severity and Mortality: a Single-center, Unblinded, Prospective, Non-interventional, Observational Study
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: ZJC202304
Record Dates: First submitted 2023-05-04; First posted 2023-05-25 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Sepsis; Inflammatory Response
Keywords: sepsis; CD8+ T cell; central memory CD8+ T cell; inflammatory response
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- septic patients: patients with sepsis defined based on Sepsis 3.0 criteria within 24 hours after admission
- healthy control group: healthy adults

SUMMARY:
Sepsis is defined as a life-threatening organ dysfunction that is caused by a dysregulated host response to infection. Severe sepsis is the most common cause of death among critically ill patients in non-coronary intensive care units (ICU). Sustained excessive inflammation and immune dysfunction have been confirmed to play a key role in organ damage and early death of sepsis patients. Therefore, it is important to reduce excessive inflammatory response mediated by immune cells and pro-inflammatory cytokines in the acute phase of sepsis.

Single-cell RNA sequencing performed on both septic patients and mice suggest that changes in Tcm (CD3+ CD8+ CD44+ CD127+ CD62L+) and Tem (CD3+ CD8+ CD44+ CD127+ CD62L -) in the acute phase of sepsis may play an important role in sepsis. In addition, animal researches showed that Tcm and Tem decreased decreased continuously at 24, 48 and 72h after cecal ligation and perforation (CLP) in mice, and the adoptive transfer of Tcm , sorting from spleen of mice 24h after CLP , but not Tem improved 7-day survival rate of sepsis mice.

This observational study is aimed to investigate the quantity and proliferation of Tcm and Tem in the acute phase of sepsis and their correlation with severity level and mortality of septic patients in ICU.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-60 years old without restriction of gender, race, religion, creed or nationality; No sedative drugs with elimination half-life were used before inclusion in the study; Patients and/or their family members know and agree to participate in the trial.

Exclusion Criteria:

History of solid organ or bone marrow transplantation; Diseases that may affect immune-related indicators, such as autoimmune diseases such as rheumatoid arthritis and SLE, or hematological malignancies such as leukemia and lymphoma; Have received radiotherapy or chemotherapy within the past 30 days, or have received immunosuppressive drugs (tripterygium, mycophenolate, cyclophosphamide, FK506, etc); Pregnancy or lactation; Chronic nephrosis; Severe chronic liver disease (child-Pugh: Grade C); alcohol or opioid dependence, mental illness, or severe cognitive impairment; Patients and/or their family members refuse to participate in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with sepsis defined based on Sepsis 3.0 criteria
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-11-03 (Actual); Study Completion 2024-11-03 (Actual)

PRIMARY OUTCOMES:
Absolute number of CD8+T subsets in the peripheral blood (0 hour) | 0 hour after study inclusion
  CD3+ CD8+ CCR7+ CD127high CD62L+ CD27high CD45RA- cells，and CD3+ CD8+ CCR7- CD127- CD62L- CD27low CD45RA- cells
Absolute number of CD8+T subsets in the peripheral blood (24 hours) | 24 hours after study inclusion
  CD3+ CD8+ CCR7+ CD127high CD62L+ CD27high CD45RA- cells，and CD3+ CD8+ CCR7- CD127- CD62L- CD27low CD45RA- cells
Absolute number of CD8+T subsets in the peripheral blood (48 hours) | 48 hours after study inclusion
  CD3+ CD8+ CCR7+ CD127high CD62L+ CD27high CD45RA- cells，and CD3+ CD8+ CCR7- CD127- CD62L- CD27low CD45RA- cells
Absolute number of CD8+T subsets in the peripheral blood (72 hours) | 72 hours after study inclusion
  CD3+ CD8+ CCR7+ CD127high CD62L+ CD27high CD45RA- cells，and CD3+ CD8+ CCR7- CD127- CD62L- CD27low CD45RA- cells
proliferation of CD8+T subsets in the peripheral blood (0 hour) | 0 hour after study inclusion
  expression of Ki67 in Tcm and Tem
proliferation of CD8+T subsets in the peripheral blood (24 hours) | 24 hours after study inclusion
  expression of Ki67 in Tcm and Tem
proliferation of CD8+T subsets in the peripheral blood (48 hours) | 48 hours after study inclusion
  expression of Ki67 in Tcm and Tem
proliferation of CD8+T subsets in the peripheral blood (72 hours) | 72 hours after study inclusion
  expression of Ki67 in Tcm and Tem
ICU length of stay | up to 4 weeks
  Length of stay in the ICU
PD-1 expression of CD8+T subsets in the peripheral blood (24 hours) | 24 hours after study inclusion
  expression of PD-1 in Tcm and Tem

SECONDARY OUTCOMES:
Mechanical ventilation time after inclusion | up to 4 weeks
  Patients requiring mechanical ventilation after study inclusion
Total hospital length of stay | up to 4 weeks
  Total length of hospital stay
In-hospital mortality | up to 4 weeks
  Mortality rates for the entire period of hospitalization
90-day readmission rate | up to 4 weeks
  Percentage of readmission to hospital within 90 days of study inclusion
Infection complications | up to 4 weeks
  Pulmonary infection, urinary tract infection, bloodstream infections, etc
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 0h after study inclusion
  0-67, higher scores correspond to more severe disease and a higher risk of death
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 24 hours after study inclusion
  0-67, higher scores correspond to more severe disease and a higher risk of death
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 48 hours after study inclusion
  0-67, higher scores correspond to more severe disease and a higher risk of death
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 72 hours after study inclusion
  0-67, higher scores correspond to more severe disease and a higher risk of death
Sequential organ failure assessment (SOFA) score | 0 hour after study inclusion
  0-43, higher scores correspond to more severe sepsis
Sequential organ failure assessment (SOFA) score | 24 hours after study inclusion
  0-43, higher scores correspond to more severe sepsis
Sequential organ failure assessment (SOFA) score | 48 hours after study inclusion
  0-43, higher scores correspond to more severe sepsis
Sequential organ failure assessment (SOFA) score | 72 hours after study inclusion
  0-43, higher scores correspond to more severe sepsis
Plasma cytokine levels | 0 hour after study inclusion
  IL-2、IL-4、IL-6、IL-10、IL-17A、IFN-γ、TNF-α
Plasma cytokine levels | 24 hours after study inclusion
  IL-2、IL-4、IL-6、IL-10、IL-17A、IFN-γ、TNF-α
Plasma cytokine levels | 48 hours after study inclusion
  IL-2、IL-4、IL-6、IL-10、IL-17A、IFN-γ、TNF-α
Plasma cytokine levels | 72 hours after study inclusion
  IL-2、IL-4、IL-6、IL-10、IL-17A、IFN-γ、TNF-α

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No